CLINICAL TRIAL: NCT03922464
Title: A Prospective, Multicenter Trial on the Efficacy and Safety of Poly-L-lactic Acid (Sculptra® Aesthetic) for the Treatment of Contour Deformities of the Buttocks Region
Brief Title: Efficacy and Safety of Poly-L-lactic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018EI - S01
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Buttock Contouring; Buttock Lifting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Poly-L-lactic acid (Sculptra® Aesthetic) — Sculptra® Aesthetic is a commercially available product that is licensed for sale in Canada. It is an injectable implant that contains microparticles of poly-L-lactic acid (PLLA), a biocompatible, biodegradable, synthetic polymer from the alpha-hydroxy-acid family. Sculptra® Aesthetic is suitable for increasing the volume of depressed areas, particularly to correct skin depressions, such as in skin creases, wrinkles, folds, scars and for skin aging. Sculptra® Aesthetic is also suitable for large volume corrections of the signs of facial fat loss (lipoatrophy).
  The safety and efficacy of Sculptra® Aesthetic has been investigated in the literature and is generally considered safe and effective. PLLA has been used successfully to reverse HIV-associated lipoatrophy as well as to rejuvenate the face, neck, décolletage, hands, abdomen and gluteal regions.

SUMMARY:
This is a phase IV prospective, multicentre, single cohort, open-label clinical trial evaluating the efficacy and safety of Poly-L-lactic acid (Sculptra® Aesthetic) for the treatment of contour deformities of the buttocks region

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Age between 30 and 60 years;
3. Indication for treatment of bilateral contour deformities;
4. Mild to moderate flaccidity in the area to be treated, according to investigator's assessment;
5. An intact immune system, as the bio-stimulatory effect of Sculptra® Aesthetic is dependent on the host response. An intact immune system, as the bio-stimulatory effect of Sculptra® Aesthetic is dependent on the host response. Immune function will be evaluated through clinical history. Exclusions will consist of both primary (genetic) and secondary (acquired) immune deficiencies. Examples include: HIV/AIDS, chemotherapy, cancers (e.g., leukemia and lymphoma), certain autoimmune diseases (e.g., myasthenia gravis, systemic lupus erythematosus), certain medications (e.g., corticosteroids, tumor necrosis factor inhibitors, anticonvulsants), and certain chronic or congenital diseases. Any type of comorbidity or clinical condition will be reviewed at the investigator's discretion.
6. . Subjects who understood and signed the Informed Consent Form (ICF) when entering the study, before performing any investigational procedure.

Exclusion Criteria:

1. Prior (i.e., <1 year) or planned use (for the duration of the study period) any other aesthetic treatment in the buttock region, such as radiofrequency, cryolipolysis, dermal subscision, plastic surgery, laser treatment, chemical peeling or any other procedure based on active dermal response;
2. Any type of comorbidity or clinical condition that, at investigator's discretion, could interfere with study assessments;
3. Using or planning to initiate restrictive diets (at investigator's discretion);
4. Using or planning to initiate use of supplements for weight loss;
5. Diabetes mellitus type 1 or type 2;
6. Autoimmune diseases, collagenosis, decompensated endocrine diseases or any disease that, at investigator's discretion, could interfere with study assessments;
7. Using or have used within the previous 3 months drugs such as corticosteroids, immunosuppressants, anticoagulants or other collagen-production inhibitors;
8. Initiated use of hormones or change in dose of hormonal replacement therapy within 3 months;
9. Practices regularly or intend to practice during the study high-performance or impact physical activities, such as weight lifting, marathon, triathlon;
10. Pregnant or breastfeeding, or wishes to get pregnant within the next 18 months, or refuses to use appropriate contraceptive method (in case of women of childbearing potential);
11. Sculptra® Aesthetic should not be used in any person who has hypersensitivity to any of the components of the product;
12. Active skin inflammation or infection in or near the treatment area;
13. Sculptra® Aesthetic should not be used in patients with known history of or susceptibility to keloid formation or hypertrophic scarring;
14. Sculptra® Aesthetic should not be used in patients with implants in the treated regions;
15. Possessing any of the contraindications for use of Sculptra® Aesthetic.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female gender.
Enrollment: 30 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-03-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects to achieve a one-point increase or higher since Baseline, on the Global Aesthetic Improvement Scale (GAIS) at Visit 6 | Month 6

SECONDARY OUTCOMES:
Assessment of adverse events (AEs) at all study visits (Visits 0-6). The incidence, seriousness, severity and relationship with the medical device of AEs reported will be evaluated. | All visits, Baseline to Month 6

OTHER OUTCOMES:
Skin hydration as measured by the corneometer | All Visits; Baseline to month 6
  The Corneometer® CM 825 will be used to measure the skin's hydration, in the center of each four buttock quadrant, at all visits.
Corporeal contour as measured by the VisioScan | All Visits; Baseline to month 6
  Evaluation of corporeal contour will be performed at all visits using The Visioscan® VC 98 to identify select, major surface irregularities and/or textural depressions caused by skin sagging (often mistaken for "cellulite").
Skin elasticity as measured by the cutometer | All Visits; Baseline to month 6
  Evaluation of corporeal contour and skin parameters, using The Cutometer® Dual Multi-Probe Adapter (MPA) 580 to measure skin's elasticity, at all visits.
cellulite severity as evaluated by the Nürnberger-Müller Scale for Cellulite | Baseline and month 3; Baseline and month 6
  Evaluations of the blinded reviewer's Nürnberger-Müller Scale for Cellulite between Baseline (Visit 0/1) and Follow up visits (Visits 4 to 6).
  The Nurnberger-Muller Scale classifies cellulite into four categories:
  Stage Zero No dimpling is seen on the skin when you are standing naked in front of the mirror. When the skin is pinched no orange peel effect is seen.
  Stage One No dimpling is seen on the skin when you are standing, but when you pinch your skin you have bumps and lumps.
  Stage two You can see dimpling or the orange peel appearance when standing naked in front of the mirror, but not when lie down.
  Stage three You can see dimpling both when you are standing and lying down.
Evaluations of patient satisfaction using the Patient Satisfaction Questionnaire at all visits | All Visits; Baseline to month 6
  The Patient Satisfaction Questionnaire is a 5-point likert scale, including:
  Very dissatisfied; Dissatisfied; Slightly satisfied; Satisfied; Very satisfied.
Evaluations of the investigator assessed GAIS scale at all visits (0-6). | Baseline to Month 6
  The Global Aesthetic Improvement Scale (GAIS) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator. The rating categories are "worse," "no change," "improved," "much improved," and "very much improved."

CONTACTS AND LOCATIONS:
Locations (1):
- Erevna Innovations Inc, Westmount, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No